CLINICAL TRIAL: NCT03870061
Title: Randomized Evaluation of a Conditional Cash Transfer Program for Routine Immunizations of Infants in Nigeria
Brief Title: Evaluation of an Infant Immunization Encouragement Program in Nigeria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GiveWell (Other)
Collaborators: New Incentives (Unknown); All Babies are Equal Initiative (Unknown)
Responsible Party: Principal Investigator, Zack Devlin-Foltz, Manager, IDinsight
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 001
Record Dates: First submitted 2019-03-04; First posted 2019-03-11 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Tuberculosis; Diphtheria; Tetanus; Pertussis; Hepatitis B; Haemophilus Influenzae Type b Infection; Pneumonia, Bacterial; Measles; Rotavirus Infections; Polio; Yellow Fever
Keywords: Randomized Controlled Trial; Vaccinations; Nigeria; Conditional Cash Transfers; Cash Incentives; Infants; Impact Evaluation; Immunization
MeSH Terms: conditions — Tuberculosis; Diphtheria; Tetanus; Whooping Cough; Hepatitis B; Haemophilus Infections; Pneumonia, Bacterial; Measles; Rotavirus Infections; Poliomyelitis; Yellow Fever

STUDY DESIGN:
Intervention Model Description: The study will be structured as a two-arm cluster RCT. One arm (83 clinics) will serve as the control and will operate as the status quo, while the other arm (84 clinics) will receive New Incentives full program. This design will measure the causal effect of New Incentives' program on the likelihood of an infant receiving a vaccine.
  New Incentives, an international non-governmental organization (NGO), is addressing the apparent shortfall in demand for immunization by offering cash incentives to caregivers for bringing their child to clinics for the first five visits of the Nigerian Routine Immunization schedule. To be eligible, the child must reside in the catchment area of the clinic and fall within the age range targeted for the vaccination in question. Infants do not need to have received the previous vaccine in the schedule to be eligible. Incentives are paid in cash by a New Incentives staff member who also ensures the infant meets the eligibility criteria outlined above.
Masking Description: Potential participants in treatment communities likely interact with implementing staff (either to receive the program, or in passing). Potential participants in control communities usually only interact with data collection staff. They are informed about the studies' general goals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Treatment (Experimental): This arm receives the full New Incentives' conditional cash transfer program (All Babies Are Equal Initiative).
  Interventions: Behavioral: All Babies Are Equal Initiative (conditional cash transfer program)

INTERVENTIONS:
Behavioral: All Babies Are Equal Initiative (conditional cash transfer program) — New Incentives, an NGO, offers cash incentives to caregivers for bringing their child to clinics for the first five visits of the Nigerian Routine Immunization schedule. These small cash transfers can provide some material benefit to new caregivers from poor communities. At a minimum, they help offset time and transport costs. The following vaccines are directly incentivized by the New Incentives' program: tuberculosis (BCG vaccine); diphtheria, tetanus, pertussis, hepatitis B and Haemophilus influenzae Type B (Pentavalent Vaccine), pneumococcal bacteria (PCV vaccine), measles vaccine.
  Arms: Treatment

SUMMARY:
Previous studies have shown that a small incentive can have a large impact on health behaviors like vaccinating children. New Incentives, an international non-governmental organization (NGO), aims to boost demand for immunization by offering cash incentives to caregivers who have their child vaccinated at a program clinic. In collaboration with New Incentives, IDinsight is conducting a study to see whether this approach will increase immunization in North West Nigeria. This study aims to investigate whether giving cash to caregivers in North West Nigeria who bring their infants to receive vaccination against common infections (tuberculosis, diphtheria, tetanus, pertussis, hepatitis B virus (HBV) infection, Haemophilus influenzae Type B (Hib), pneumococcal bacteria, measles, rotavirus, polio, yellow fever) increases the proportion of children who are immunized. The study's main hypothesis is that New Incentives' program will increase the percentage of children immunized with BCG, any PENTA, or Measles 1 by an average increase of at least 7-percentage points across all program clinics that share a similar profile to the clinics New Incentives will operate in at scale. The study is taking place in Jigawa, Katsina, and Zamfara States between August 2017 and January 2020.

DETAILED DESCRIPTION:
The study will be structured as a two-arm cluster RCT with clinics catchment areas as clusters. One arm will serve as the control (83 clinics) and will operate as the status quo, while the other arm will receive New Incentives' full program (84 clinics). This design will measure the causal effect of New Incentives' program on the likelihood of an infant receiving a vaccine. The unit of treatment and randomization is the clinic catchment, while the unit of measurement for the key outcomes is the individual infant.

Eligible caregivers who bring their infant(s) to a treatment group health facility for immunizations are first enrolled in the program by New Incentives staff, who record caregiver and infant details. If the child has received the vaccination, the caregiver receives the cash incentive, and instructions on when to return for the next vaccination and incentive payment.

Data collection of outcome measures takes place at three points (baseline, midline, and endline) using a series of self-reported surveys of caregivers, examination of the child's health card (where available) and reviewing clinic records. Baseline was completed between August and October 2017, midline is scheduled for March 2019, and endline is planned for November 2019 to January 2020. Across all outcome measurements, sampled infants will be aged between 12 and 16 months (though baseline surveyed some infants aged up to 24 months to increase sample size). These age groups are sampled as they are well beyond the age at which children should receive the program vaccinations. (The Nigerian Routine Immunization schedule aims to give the program vaccinations between birth and 9 months old.) IDinsight does not follow the same infants from baseline to midline to endline but, rather, compares coverage rates in the same age group at each point in time. From the perspective of the participant, taking part in the study involves receiving a researcher into their home, providing informed consent, and answering a 1-hour survey.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0 to 16 months can be enrolled in the program and incentives paid to their caregivers
* Children aged 12 to 16 months will have their data measured at endline
* All participants must reside in study clinic catchment areas.
* Vaccination status will be measured by caregiver survey. Caregivers must consent to the survey

Exclusion Criteria:

* Residence outside the study area (self-reported)
* Outside the age range (self-reported)

Ages: 12 Months to 16 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5187 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
The probability that a 12- to 16-month-old in a community served by a study clinic received BCG (based on caregivers' report of their child's vaccination history) | 12 to 16 months after birth
The probability that a 12- to 16-month-old in a community served by a study clinic received at least one dose of PENTA (based on caregivers' report of their child's vaccination history) | 12 to 16 months after birth
The probability that a 12- to 16-month-old in a community served by a study clinic received Measles 1 (based on caregivers' report of their child's vaccination history) | 12 to 16 months after birth

SECONDARY OUTCOMES:
The probability that a 12- to 16-month-old in a community served by a study clinic is fully immunized (loose and strict) (based on caregivers' report of their child's vaccination history) | 12 to 16 months after birth
The timeliness of vaccination, particularly for Measles 1, among 12- to 16-month-olds in communities served by a study clinic (based on caregivers' report of their child's vaccination history) | 12 to 16 months after birth
The average number of vaccines received per 12- to 16-month-old child in communities served by a study clinic (based on caregivers' report of their child's vaccination history) | 12 to 16 months after birth
The percentage of 12- to 16-month-olds in communities served by a study clinic who received at least one injectable vaccine (based on caregivers' report of their child's vaccination history) | 12 to 16 months after birth
The probability that a 12 to 16-month old in a community served by a study clinic received at least one dose of PCV? | 12 to 16 months after birth
The change over time in the volume of BCG, Penta 1, Penta 2, Penta 3, and Measles vaccinations recorded in clinic administrative records between treatment and control | 12 to 16 months after birth

CONTACTS AND LOCATIONS:
Overall Officials: Alison Connor, PhD, Study Director — IDinsight
Locations (3):
- Nigeria (3):
  - Primary Health Care facilities across Jigawa State, Various Cities, Jigawa State
  - Primary Health Care facilities across Katsina State, Various Cities, Katsina State
  - Primary Health Care facilities across the Zamfara State, Various Cities, Zamfara State

IPD SHARING:
Plan to Share IPD: Undecided
All participant-level data is anonymized through removing any information that could lead to back-tracking the identity of the respondent - each respondent is allocated a random identification number in place of their name. Anonymized data are currently stored in a password-protected repository on IDinsight's Dropbox site. Access is restricted to IDinsight staff that are on the project.
  IDinsight and New Incentives collect various clinic-level data as well for use as covariates and to inform operational decisions. These data are stored in the same repositories and in New Incentives' own password-protected internal dashboard.
  Requests for access to data can be made directly to IDinsight (Manager: Zack Devlin-Foltz (zack.devlinfoltz@idinsight.org) and Corresponding Investigator: Dr. Niklas Heusch (niklas.heusch@idinsight.org))

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-29): https://cdn.clinicaltrials.gov/large-docs/61/NCT03870061/Prot_SAP_001.pdf